CLINICAL TRIAL: NCT02708992
Title: The Pharmacokinetics of Extended Duration High-Dose Cefixime Co-administered With Azithromycin for the Decreased Susceptibility of Neisseria Gonorrhoeae: A Phase I Pilot Study
Brief Title: Cefixime / Azithromycin pK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-0031; HHSN272201500006I
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-07-19

CONDITIONS: Gonorrhoea
Keywords: Azithromycin; Cefixime; Duration; High-Dose; Neisseria gonorrhoeae; Pharmacokinetics; Susceptibility
MeSH Terms: conditions — Gonorrhea; Disease Susceptibility | interventions — Azithromycin; Cefixime

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cefixime/Azithromycin (Experimental): Eight participants will receive three oral doses of 800 mg cefixime (q 8 hours) on Day 1, followed by three oral doses of 800 mg cefixime (q 8 hours)+ one oral dose of 1000 mg azithromycin (with first dose of cefixime) on day 10
  Interventions: Drug: Azithromycin; Drug: Cefixime

INTERVENTIONS:
Drug: Azithromycin
Drug: Cefixime

SUMMARY:
This is a PK study of a multi-dose oral cefixime regimen (three 800 mg doses given on a q 8-hour schedule) alone and also co administered with a single 1000 mg oral dose of azithromycin, both within a 24-hour period, in order to achieve total serum cefixime levels of mcg/mL for at least 20 hours. This will determine the tolerability of the regimen and whether there are significant changes in cefixime PK after co-administration. The primary pharmacokinetic objectives are: to determine if a cefixime dosing regimen of three 800 mg doses given alone, on a q 8-hour schedule achieves a total serum cefixime level that exceeds 2.0 mcg/mL for at least 20 hours; to determine if a cefixime dosing regimen of three 800 mg doses given on a q 8 hour schedule co-administered with a single 1000 mg of azithromycin, achieves a total serum cefixime level that exceeds 2.0 mcg/mL for at least 20 hours; and to evaluate whether a single 1000 mg dose of azithromycin alters the PK of a three dose regimen of 800

DETAILED DESCRIPTION:
This is a PK study of a multi-dose oral cefixime regimen (three 800 mg doses given on a q 8-hour schedule) alone and also co administered with a single 1000 mg oral dose of azithromycin, both within a 24-hour period, in order to achieve total serum cefixime levels of mcg/mL for at least 20 hours. This will determine the tolerability of the regimen and whether there are significant changes in cefixime PK after co-administration. The primary pharmacokinetic objectives are: to determine if a cefixime dosing regimen of three 800 mg doses given alone, on a q 8-hour schedule achieves a total serum cefixime level that exceeds 2.0 mcg/mL for at least 20 hours; to determine if a cefixime dosing regimen of three 800 mg doses given on a q 8 hour schedule co-administered with a single 1000 mg of azithromycin, achieves a total serum cefixime level that exceeds 2.0 mcg/mL for at least 20 hours; and to evaluate whether a single 1000 mg dose of azithromycin alters the PK of a three dose regimen of 800 mg cefixime given on a q 8-hour schedule. The primary safety objectives are to assess the safety and tolerability of a treatment regimen that includes three doses of 800 mg cefixime; to assess the safety and tolerability of a treatment regimen that includes three doses of 800 mg cefixime co-administered with a single 1000 mg dose of azithromycin. The study will take place for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects between 18 and 45 years, inclusive 2. Ability to understand the consent process and procedures 3. Informed consent obtained and signed prior to initiation of any study procedures 4. Subjects agree to be available for all study visits 5. Negative breathalyzer for alcohol 6. Agreement by female subjects with reproductive potential to use an adequate method of contraception during the study and for 30 days after last study drug administration. Female subjects must agree to the use of TWO reliable methods of contraception while receiving study drug and for 30 days after last study drug administration if sexually active, which can include: condoms, spermicidal gel, diaphragm, hormonal or non-hormonal intrauterine device, surgical sterilization, oral contraceptive pill (OCP), and depot progesterone injections.

Exclusion Criteria:

1. Subjects who take any prescription medication on a regular basis (except OCPs), including but not limited to, anti-psychotics, anti-depressants, anti-epileptics, cardiac medications, and antihypertensives. 2. Subjects who take any OTC drugs or herbal remedies on a regular basis, especially those that have been associated with a risk of QT prolongation such as antiemetics (ondansetron, granisetron, dolasetron, hydroxyzine), antihistamines (terfenadine, astemizole, hydroxyzine, diphenhydramine), GI stimulants (cisapride, domperidone, metoclopramide), and homeopathic agents (cinchona, licorice extract- glycyrrhizin). 3. Hypertension with confirmed systolic blood pressure >140 mmHg or confirmed diastolic blood pressure > 90 mmHg, measured after 10 to 15 minutes of rest 4. Morbid obesity (BMI >/= 35 kg/m^2) 5. Current diagnosis of pulmonary disease 6. History or current diagnosis of diabetes 7. Autoimmune disorders, such as lupus, Wegener's, rheumatoid arthritis 8. History of malignancy except low-grade skin cancer, (i.e., basal cell carcinoma thought to be cured) 9. Known diagnosis of prolonged QT interval, congenital long QT syndrome, bradyarrhythmias or uncompensated heart failure 10. History of alcohol abuse 11. History of seizure disorder 12. History of renal disease 13. Chronic renal, hepatic, or pulmonary disease or other condition that could interfere with the absorption of the study drug or predispose to adverse GI events (e.g., surgical resection of significant proportions of the stomach or bowel, gastric bypass, gastric banding, irritable bowel syndrome, inflammatory bowel disease) 14. Positive serology results for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies 15. Subjects who have taken any prescription drugs in the previous 14 days or within five half-lives before dosing 16. Ingestion of OTC medications or herbal supplements within seven days of dosing 17. Positive urine drug screen for marijuana, cocaine, amphetamines, opiates, phencyclidine, barbiturates, or benzodiazepines 18. History of allergic reaction or intolerance to cephalosporins 19. History of allergic reaction to penicillin (all stages) 20. History of allergic reaction to azithromycin, erythromycin, or any macrolide or ketolide antibiotic 21. History of jaundice or hepatic dysfunction associated with prior use of azithromycin 22. Males with a QTcF > 430ms or Females with a QTcF >450ms (Fridericia's correction) on screening 23. Positive pregnancy test; pregnant or nursing women 24. Screening laboratory tests > Grade 1 as defined by Appendix B 25. Any specific condition that, in the judgment of the Investigator, precludes participation because it could affect subject safety.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
AUC from 0 to infinity [AUC0-infinity] | Day 1,2,3,10,11,12 and at early termination
Averaged composite plasma cefixime levels will be used to generate PK curves of cefixime levels versus time | Day 1,2,3,10,11,12 and at early termination
Elimination half-life (t1/2) | Day 1,2,3,10,11,12 and at early termination
Elimination rate (lambda z) | Day 1,2,3,10,11,12 and at early termination
Individual plasma cefixime levels will be used to generate PK curves of cefixime levels versus time | Day 1,2,3,10,11,12 and at early termination
Peak cefixime level (Cmax) | Day 1,2,3,10,11,12 and at early termination
Safety blood test results | Day: -28,-1, 2, 3, 9, 11, 12, 17 and at early termination
Safety urinanalysis results | Day: -28, -1, 2, 3, 9, 11, 12, 17 and at early termination
Subject reported AEs | Day: 1, 2, 3, 9, 10, 11, 12, 17 and at early termination
Subject reported serious adverse events (SAEs) | Day: 1, 2, 3, 9, 10, 11, 12, 17 and at early termination
Targeted clinical evaluations | Day: -1,1, 2, 3, 9, 10, 11, 12, 17 and at early termination
Time that cefixime levels exceed four times the MIC of 0.5 mcg/mL (i.e., a plasma level of 2.0 mcg/mL) | Day 1,2,3,10,11,12 and at early termination
Time to peak drug level (Tmax) | Day 1,2,3,10,11,12 and at early termination
Total area under the curve (AUC from 0 hours to the time of next dosing [AUC0-t]) | Day 1,2,3,10,11,12 and at early termination
Total plasma concentrations of cefixime | Day 1,2,3,10,11,12 and at early termination

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University School of Medicine - Duke Clinical Research Institute - Duke Clinical Research Unit, Durham, North Carolina, United States